CLINICAL TRIAL: NCT03445793
Title: : TRANSITION: An Observational Study of the Effects on Sweat Chloride and Clinical Outcomes of Transition From Lumacaftor/Ivacaftor to Tezacaftor/Ivacaftor (Tez/Iva)
Brief Title: : TRANSITION: An Observational Study of Transition From Lumacaftor/Ivacaftor to Tezacaftor/Ivacaftor (Tez/Iva)
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Jennifer Taylor-Cousar, MD, Principal Investigator, Co-Director/CF TDN Director, Adult CF Program, National Jewish Health
Other Study IDs: HS-3145
Record Dates: First submitted 2018-02-05; First posted 2018-02-26 (Actual); Results first posted 2021-10-01 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis (CF)
Keywords: DeltaF508deletion (F508del) mutation in 2 copies
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single center study of clinical and laboratory outcomes in patients ≥ 12 who transition from use of Orkambi to tez/iva. Clinical and laboratory measurements will be measured at baseline, 1 month, 3 months, and 6 months after initiation of tez/iva. Change from baseline at 6 months pre-specified will be reported. The length of study participation will be approximately 6 months.

DETAILED DESCRIPTION:
While cystic fibrosis (CF) therapeutic development previously targeted the signs and symptoms of the disease, in the last 5 years, two drugs that treat the basic defect in CF have been approved, ivacaftor (iva) and lumacaftor/ivacaftor (lum/iva). This class of drugs, deemed cystic fibrosis transmembrane conductance regulator (CFTR) modulators, variably improve CFTR function as measured by pilocarpine iontophoresis and sweat collection, and clinical outcomes including lung function, body mass index (BMI), rate of exacerbations and patient reported quality of life.

In patients with the G551D mutation who received iva, there was a marked decrease in sweat chloride and marked improvement in lung function as measured by absolute change from baseline of percent predicted expiratory volume in 1 second (ppFEV1). The clinical outcomes assessed in the phase III studies of lum/iva and tez/iva were similar, and included lung function, rate of pulmonary exacerbations, BMI, and CFQ-R scores. While the correlation between improvement in sweat chloride and lung function is poor, and a minimum threshold for change in sweat chloride that correlates with clinical outcomes has yet to be defined, it has also not been determined if an increase in sweat chloride caused by a transition from one drug to another would adversely impact clinical outcomes. Outcomes between the phase III studies of lum/iva and tez/iva were similar, tez/iva has three advantages that are likely to make it more appealing to patients and providers than lum/iva including positive clinical efficacy data, fewer drug-drug interactions, and an improved tolerance profile.

Following tez/iva approval, a rapid uptake of tez/iva for patients homozygous for F508del CFTR is expected; as a result of the transition from lum/iva to tez/iva, sweat chloride will increase possibly resulting in an adverse impact on clinical outcomes. This study aims to determine the rationale for patient transition from lum/iva to tez/iva, in addition to evaluate the impact of transition on CFTR function, pulmonary health, gastrointestinal health, and general health. While it is possible that there will be no change in sweat chloride or small changes that are without clinical significance, systematic collection of data as patients transition from lum/iva to tez/iva would permit rapid identification of any safety issues. Because the U.S. always leads the way with approval and reimbursement of new therapeutics, our experience with this transition will help guide its conduct for physicians and patients in the rest of the world.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Male or female subjects greater than or equal to 12 years of age
* Ability to reproducibly perform spirometry testing
* Physician decision to treat with tezacaftor/ivacaftor (Smydeko)
* Ability to understand and sign a written informed consent or assent and comply with the requirements of the study
* Continuous use of orkambi for at least 1 month prior to visit 1

Exclusion Criteria:

* History of hypersensitivity to tezacaftor and/or ivacaftor
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Any acute lower respiratory symptoms treated with oral, inhaled or intravenous antibiotics (IV) or systemic corticosteroids within the 2 weeks prior to Visit 1
* Major or traumatic surgery within 12 weeks prior to Visit 1
* For women of child-bearing potential: a positive pregnancy test at Visit 1
* Unable or unwilling to fast (including no enteric tube feedings) for at least 6 hours prior each visit
* Initiation of any new chronic therapy within 4 weeks prior to Visit 1
* Use of an investigational agent within 28 days prior to Visit 1
* Use of chronic oral corticosteroids within 28 days prior to Visit 1
* Treatment for nontuberculous mycobacterial (NTM) infection, consisting of greater than or equal to two antibiotics (oral, IV, and/or inhaled) within 28 days prior to Visit 1
* History of lung or liver transplantation, or listing for organ transplantation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis with 2 copies of F508del mutation.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Taylor-Cousar, MD, MSCS, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Heatlh, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center recruitment from March 2018 until November 2019.
Pre-assignment Details: Participant must complete baseline visit while on lumacaftor/ivacaftor prior to transition to tezacaftor/ivacaftor.
Groups:
- Observational: Participants who have cystic fibrosis and are clinically stable at time of transition from Lumacaftor/Ivacaftor to tezacaftor/ivacaftor as a continuous treatment as determined by their clinical physician.
Period: Overall Study
Arm/Group | Observational
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Observational
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of consent
  years | 28.4 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Cystic Fibrosis Mutation Type [Count of Participants; unit: Participants]
  Homozygous for F508del | 5
  Heterozygous for F508del | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.3 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sweat Chloride Concentration in Millimoles/Liter From Baseline at 6 Months Pre-specified to be Reported
Description: Sweat chloride is a measure of cystic fibrosis transmembrane conductance regulator function. The calculations represent the average change from baseline to the average change at 6 months.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Observational
Number analyzed (Participants) | 5
mmol/L | 10.2 [-12.1 to 32.5]

2. Secondary Outcome: Rationale for Transition Per Physician Questionnaire
Description: Questionnaire to determine the treating physician's reason for transition to tezacaftor/ivacaftor from lumacaftor/ivacaftor
Time Frame: 1 day (the questionnaire is done once at visit 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 5
Participants
  Side Effects/Intolerance of Orkambi | 4
  No benefit on Orkambi | 1

3. Secondary Outcome: Rationale for Transition Per Subject Questionnaire
Description: Questionnaire to determine the subject's reason for transition to tezacaftor/ivacaftor from lumacaftor/ivacaftor
Time Frame: 1 day (the questionnaire is done once at visit 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 5
Participants
  "Orkambi is no longer working for me" | 1
  No benefit on Orkambi | 1
  Side effects/Intolerance on Orkambi | 2
  Personal desire to try new therapy | 1

4. Secondary Outcome: Pulmonary Exacerbations
Description: Number of pulmonary exacerbations requiring oral or IV antibiotics
Time Frame: One year prior to study entry (time of consent) and during study participation
Measure: Mean (Standard Deviation); unit: Pulmonary Exacerbations
Arm/Group | Observational
Number analyzed (Participants) | 5
Pulmonary Exacerbations | 3.2 (3.96)

5. Secondary Outcome: Change in Percent Predicted (ppFEV1) Value From Baseline at 6 Months Pre-specified to be Reported
Description: Pulmonary function by spirometry, percent predicted forced expiratory volume in 1 second. The calculations represent the average change from baseline to the average change at 6 months.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: percent predicted (ppFEV1)
Arm/Group | Observational
Number analyzed (Participants) | 5
percent predicted (ppFEV1) | -2.0 [-5.93 to 1.93]

6. Secondary Outcome: Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score From Baseline at 6 Months
Description: CF-related quality of life measure is a validated, CF specific, patient reported outcome (PRO). This portion of the PRO is specific to respiratory symptoms. The scaled score for each domain ranges from 0 (worst condition) to 100 (best condition), with higher scores indicating better health in respiratory domain.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Observational
Number analyzed (Participants) | 5
score on a scale | -11.3 [-25.9 to 3.2]

7. Secondary Outcome: Change in Weight in Kilograms From Baseline at 6 Months Pre-specified to be Reported
Description: Weight is a reflection of nutrition status in CF and is expected to improve with CFTR modulation. The calculations represent the average change from baseline to the average change at 6 months.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Observational
Number analyzed (Participants) | 5
kg | 2.0 (2.68)

8. Secondary Outcome: Change in BMI in kg/m^2 From Baseline at 6 Months Pre-specified to be Reported
Description: BMI is a reflection of nutrition status in CF and is expected to improve with CFTR modulation. The calculations represent the average change from baseline to the average change at 6 months.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Observational
Number analyzed (Participants) | 5
kg/m^2 | -0.67 [-1.83 to 0.48]

9. Secondary Outcome: Number of People With Undetectable or Normal Fecal Elastase Measurements at 6 Months Pre-specified to be Reported
Description: Fecal elastase in micrograms/gram. Fecal elastase is a measure of pancreatic function: Less than 100 mcg/g indicates severe exocrine pancreatic insufficiency, 100-200 mcg/g indicates moderate to mild insufficiency, greater than 200 indicates normal pancreatic function. The count represents the number of participants with either an undetectable fecal elastase level or normal level at 6 months, indicating change in pancreatic function at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational
Number analyzed (Participants) | 5
Participants
  Undetectable <15 | 5
  Normal Result | 0

10. Secondary Outcome: Change in Gastrointestinal Symptom Tracker Score From Baseline to 6 Months
Description: The Exocrine Pancreatic Insufficiency (EPI) GI Symptom Tracker is meant to measure the impact treatment is having on GI symptoms, perceived by person completing the tracker. Participants answer 24 symptom questions on a scale from almost always to never (scale 4 to 1). Higher scores reflect more challenges/problems related to GI symptoms. For purposes of this outcome measure, subscales were combined to compute a total score (minimum score 24, maximum score 96). The difference of total scores from baseline at 6 months were calculated to measure average overall change in GI symptoms.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observational
Number analyzed (Participants) | 5
units on a scale | 0.6 (8.20)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Observational
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=5)
Hospitalization due to pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (16)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=5)
Increased cough after stopping Tezacaftor/Ivacaftor (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject stopped treatment with Tezacaftor/Ivacaftor after transitioning from Lumacaftor/Ivacaftor
Exacerbation of Chronic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The limitation is the small sample size. Less patients with cystic fibrosis transitioned from lumacaftor/ivacaftor to tezacaftor/ivacaftor than expected. The enrolled number of patients left the study underpowered to detect differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT03445793/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03445793/ICF_001.pdf